CLINICAL TRIAL: NCT06575504
Title: Ultrasonographical Study of Suprarenal Gland in High Risk Neonates
Brief Title: Ultrasonographical of Suprarenal Gland in High Risk Neonates
Acronym: USSGneonates
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, safaa ELMeneza, Professor, Al-Azhar University
Other Study IDs: AlAzharU; 2462 (Other: AlAzharU)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Insuffeciency of the Suprarenal Gland
Keywords: Doppler Ultrasound; Suprarenal gland; high risk neonates; NICU

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates: High risk newborn infants admitted to NICU
  Interventions: Diagnostic Test: Ultrasonographical examination

INTERVENTIONS:
Diagnostic Test: Ultrasonographical examination — Study size and Doppler / blood flow / of the suprarenal gland

SUMMARY:
Observation study The aim is to study the suprarenal blood flow among high-risk neonates and its relation to the risk factors

DETAILED DESCRIPTION:
Ultrasonographical study of the suprarenal gland in high risk newborn infants Al-Zhrraa University hospital Sample size 105 Inclusion criteria: 1- High-risk newborn 2- Need NICU admission Exclusion criteria: Cases with Major congenital anomalies and NEC Primary outcome: Abnormal suprarenal blood flow Informed consent will be obtained from all parents and mothers of the newborns enrolled in the study.

All cases will be subjected to - Full history taking: (prenatal -natal - postnatal). According to the routine admission sheet of NICU of Alzahraa University Hospital, Faculty of Medicine for girls, AL-Azhar University, Cairo, Egypt.

Through clinical examination (APGAR score -estimation of gestational age using modified Ballard score "Ballard, 1991" - body weight - severity of respiratory illness using Downs score and Silverman's score).

Laboratory investigations:

* Blood gases.
* Serum electrolytes and blood glucose.
* CBC. CRP.
* Liver and kidney functions. Radiological evaluation: in the form of Abdominal and chest x-ray. Ultrasonographical studies were done for suprarenal gland blood flow. - Statistical Analysis, Data were collected, revised, coded, and entered into the statistical package for social science (SPSS)

ELIGIBILITY:
Inclusion Criteria:

* High risk neonates

Exclusion Criteria:

* congenital anomalies

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates with high risk illness
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Adrenocortical insufficiency | 12 months
  Blood flow velocity RI ED TMAX

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine for girls, Cairo, Pediatrics/neonatology, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Used for results publications
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2 years
Access Criteria: Journal authority
URL: https://guides.lib.umich.edu/datamanagement/clinicaltrials

REFERENCES:
- Available data/document: Study Protocol — https://guides.lib.umich.edu/datamanagement/clinicaltrials